CLINICAL TRIAL: NCT05092789
Title: Comparison of Kinesio Taping and Cervical Thrust Manipulation in Patients With Mechanical Neck Pain
Brief Title: Comparison of Kinesio Taping and Cervical Thrust Manipulation in Neck Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REC/00946 Taqdees e Maryam
Record Dates: First submitted 2021-09-17; First posted 2021-10-26 (Actual); Last update posted 2022-03-23 (Actual); Status verified 2022-03

CONDITIONS: Neck Pain
Keywords: Mechanical neck pain; Kinesio taping; Cervical manipulation
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Kinesio taping group (Experimental): Participants in this group will receive treatment through standardized therapeutic Kinesio taping along with conventional therapy.
  Tape will be water proof, porous, adhesive,with width of 5cm and thickness of 0.5 mm.
  Interventions: Other: Kinesio taping group
- Cervical thrust manipulation group (Experimental): Participants in this group will receive treatment via cervical thrust manipulation along with conventional therapy.
  Manipulation will be directed on mid cervical spine.
  Interventions: Other: Cervical thrust manipulation group
- Conventional therapy group (Active Comparator): .Participants of this group will receive only conventional therapy which will include: Hot pack for 10 minutes Stretching Exercises
  Interventions: Other: Conventional therapy group

INTERVENTIONS:
Other: Kinesio taping group — Participants in this group will receive treatment through standardised therapeutic kinesio taping along with conventional therapy.
  Tape will place over the posterior cervical extensor muscle, from insertion to the origin, with the patient's neck in cervical contralateral side-bending and rotation.
  Duration of kinesio tape will be of 48 hours with 50-100% tension.
  Participants of this group will also receive conventional therapy which will include:
  Hot pack for 10 minutes Stretching exercises of the neck muscles. This protocol is for 6 weeks. The sessions will be given twice a week making it a total of 12 sessions.
  Arms: Kinesio taping group
Other: Cervical thrust manipulation group — Participants of this group will receive treatment via cervical thrust manipulation along with conventional therapy.
  For mid cervical spine thrust manipulation, the patient will be in supine lying position,with cervical spine in neutral position.
  The therapist will cradle the patients head with the other hand. Gentle ipsilateral cervical side flexion and contralateral rotation will introduce until tension will perceive in target tissues at contact point. A high velocity, low amplitude thrust manipulation, will direct upward and medially in direction of subject's contralateral eye.
  Participants of this group will also receive conventional therapy which will include:
  Hot pack for 10 minutes Stretching exercises of the neck muscles. This intervention protocol is for 6 weeks. The sessions will be given twice a week making it a total of 12 sessions with 1 month follow up.
  Arms: Cervical thrust manipulation group
Other: Conventional therapy group — Participants of this group will receive only conventional therapy which will include:
  Hot pack for 10 minutes Stretching Exercises of neck muscles. For sternocleidomastoid stretching, the subject will ask to sit or stand facing forward, exhale and slowly turn your head to right, by keeping shoulder relaxed and down,inhale and return to the center, then turn to look at your left shoulder, ask to hold this position for 30 seconds and do 3 repetitions.
  For Trapezius stretching, patient is seated upright, therapist then passively move right ear to right shoulder.
  This study includes interventional protocol of 6 weeks. The session will be given twice a week making it a total of 12 sessions with 1 month follow up.
  Arms: Conventional therapy group

SUMMARY:
To compare the effects of kinesio taping, cervical thrust manipulation and conventional therapy on neck pain, functional status and range of motion

DETAILED DESCRIPTION:
Neck pain is most prevalent condition affecting globally, which also create threats to the individuals. Mechanical neck pain affects mainly two third of population at some time in life possibly in middle age, some people may be acute mechanical neck pain while some leading to chronic stage. Mechanical neck disorders usually associated with pain, decreased cervical mobility, spasm. Often neck pain is mechanical in nature, according to literature mechanical neck pain is defined as, that pain originating from cervical spine which may be aggravated with cervical motion, prolonged posture, muscular stiffness. Due to widespread occurrence of mechanical neck pain mainly in modern society, proper interventional strategies of this problem is needed to facilitate that problem. Incidence of neck pain may range from 10.4-23.3%in one year, while according to previous literature prevalence of neck pain was 0.4 to 86.8%, with high proportion in office workers, computer users, and females especially 35 to 55 years. Pain, stiffness, tenderness and restricted mobility is most common symptoms associated with neck pain, manual therapy techniques, exercises, mobilization, manipulations, kinesio taping are treatment strategies used for this problem may improve neck pain.

The main purpose of my study is to improve neck pain, discomfort and functional status in patients with mechanical neck pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects having mechanical neck pain.
* participants having neck pain more than 1 month.

Exclusion Criteria:

* History of serious pathology (Malignancy, inflammatory disorders).
* Cervical spinal surgery.
* History of trauma or fracture.
* Vascular syndromes.
* Neurological and cardiac pathologies.

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2021-10-26 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Cervical range of motion | 6 weeks
  This tool will be used to detect cervical range of motion like cervical flexion, cervical extension, cervical side bending and cervical rotation at the baseline and at the end of 6th week.
  Cervical spines range of motion is 80-90 degrees of flexion, 70 degrees of extension, 20-45 degrees of lateral bending and up to 90 degrees of rotations.

SECONDARY OUTCOMES:
Numerical pain rating scale | 6 weeks
  This tool will be used in order to measure the intensity of pain at the baseline and at the end of 6th week.
  Maximum score on the scale is 10. Lower score means no pain and vice versa.
  Interpretation of the scores are as following:
  0 indicates no pain. 1-3 indicates mild pain. 4-7 indicates moderate pain. 8-10 indicates worst possible pain.

OTHER OUTCOMES:
Neck functional stability | 6 weeks
  This tool will be used to measure functional stability of neck at the baseline. Maximum score on the scale is 50. Lower score means less disability of the neck and vice versa.
  Interpretation of the scores are as following:
  0-4 indicates no disability. 5-14 indicates mild disability. 15-24 indicates moderate disability. 25-34 indicates severe disability. Above 34 indicates complete disability

CONTACTS AND LOCATIONS:
Overall Officials: Saad Rauf, Master, Principal Investigator — Riphah International University
Locations (1):
- Natural Medicine and Rehabilitation Center, Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No